CLINICAL TRIAL: NCT00002334
Title: A Randomized, Multicenter, Double-Blind, Phase III, Parallel Study of Zidovudine (AZT) Alone Versus AZT Plus Zalcitabine (Dideoxycytidine; ddC) Versus AZT Plus Saquinavir Mesylate (Ro 31-8959 ; HIV Proteinase Inhibitor) Versus AZT Plus ddC Plus Ro 31-8959 in Previously Untreated or Minimally Pretreated HIV-Infected Patients With CD4 Lymphocyte Counts From 50 to <= 350 Cells/mm3
Brief Title: A Study of Zidovudine (AZT) Used Alone or in Combination With Other Anti-HIV Drugs in HIV-Infected Patients With Little or No Previous Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 229B; SV 14604C; SV 14604A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-09

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Saquinavir; HIV Protease Inhibitors
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Saquinavir; Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Saquinavir
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To compare, in zidovudine (AZT)-naive patients, the safety, tolerance, and efficacy of saquinavir mesylate (Ro 31-8959) alone versus AZT alone versus AZT in combination with Ro 31-8959, zalcitabine (ddC), or both. To compare various disease markers among the different regimens.

DETAILED DESCRIPTION:
Patients are randomized to receive a minimum of 80 weeks of AZT alone, AZT plus ddC, AZT plus Ro 31-8959, or all three drugs.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Erythropoietin and G-CSF.

Concurrent Treatment:

Allowed:

* Local skin radiotherapy.

Patients must have:

* HIV infection.
* CD4 count 50 - 350 cells/mm3.
* No prior antiretroviral therapy OR less than 16 weeks of prior AZT.
* No acute serious opportunistic infections requiring immediate treatment.
* No unexplained fever persisting for 14 days within 90 days prior to study entry.
* No significant unexplained diarrhea persisting for 14 days within 30 days prior to study entry.
* No visceral Kaposi's sarcoma or lymphoma currently requiring chemotherapy and/or radiotherapy.
* Life expectancy of at least 80 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malabsorption.
* Severe chronic diarrhea.
* Inadequate oral intake (unable to eat one or more meals daily because of chronic nausea, emesis, or abdominal/oral-esophageal discomfort).
* Any grade 3 or worse toxicity.
* Inability to comply with study requirements.

Concurrent Medication:

Excluded:

* Other investigational agents.
* Antineoplastic agents.
* Biologic response modifiers (including interferons).
* Foscarnet.
* Anti-HIV drugs other than the study drugs.

Concurrent Treatment:

Excluded:

* Radiotherapy (other than local skin radiotherapy).

Patients with the following prior condition are excluded:

History of non-Hodgkin's lymphoma.

Prior Medication:

Excluded:

* Acute therapy for opportunistic infection within 14 days prior to study entry.
* Prior HIV proteinase inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000

CONTACTS AND LOCATIONS:
Locations (26):
- United States (25):
  - Phoenix Body Positive, Phoenix, Arizona
  - UCD Med Ctr, Sacramento, California
  - Davies Med Ctr, San Francisco, California
  - Mount Zion Med Ctr / UCSF, San Francisco, California
  - Pacific Oaks Med Group, Sherman Oaks, California
  - Sunnyvale Med Clinic, Sunnyvale, California
  - Novum Inc, Washington D.C., District of Columbia
  - Howard Univ, Washington D.C., District of Columbia
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Tulane Univ Med School, New Orleans, Louisiana
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - HIV Wellness Ctr / Univ Med Ctr, Las Vegas, Nevada
  - Beth Israel Med Ctr, New York, New York
  - Harkness Pavilion, New York, New York
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Univ of Oklahoma Health Science / Pharmacy Practice, Oklahoma City, Oklahoma
  - Novum Inc, Pittsburgh, Pennsylvania
  - Respiratory Associates, Corpus Christi, Texas
  - N Texas Ctr for AIDS & Clin Rsch, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Thomas Street Clinic / Baylor College of Medicine, Houston, Texas
  - Univ of Washington, Seattle, Washington
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico

REFERENCES:
- [Background] Collier CA, Coombs RW, Schoenfeld DA, Bassett R, Hooper C, Timphone J, Baruch A, Corey L. A comparative study of saquinavir (SAQ), and zidovudine (ZDV) vs. ZDV and zalcitabine (ddC) vs. SAQ, ZDV, and ddC. Program Abstr Intersci Conf Antimicrob Agents Chemother. 1994 Oct 4-7:60